CLINICAL TRIAL: NCT00663299
Title: COMPLEX Post Market Surveillance Electronic Registry
Acronym: COMPLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 03-2004
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Intracranial Aneurysm
Keywords: Intracranial aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trufill Detachable Coil System (Other): There is only one treatment arm in the registry and it is all patients receiving treatment with Trufill Detachable Coil System. The use of bare platinum coils for the endovascular occlusion of cerebral aneurysms.
  Interventions: Device: Endovascular Embolization Device

INTERVENTIONS:
Device: Endovascular Embolization Device — The TRUFILL DCS and TRUFILL DCS ORBIT Detachable Coils are each an embolic coil system that consists of a platinum detachable coil, a delivery system (delivery tube and coil introducer) and a syringe. Each system has been designed to deliver, position and detach embolic coils in order to embolize intracranial aneurysms
  Other Names: TRUFILL® DCS and TRUFILL DCS ORBIT Detachable Coils

SUMMARY:
To demonstrate performance of TRUFILL DCS and TRUFILL DCS ORBIT Detachable Coils in the treatment of aneurysms.

DETAILED DESCRIPTION:
This Post Market Surveillance Registry collect baseline characteristics, aneurysmal features, procedural and follow-up information, and complications/adverse events on the performance intracranial aneurysms treated with the Trufill DCS Orbit detachable platinum coils.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with angiographically documented aneurysms,
2. Either ruptured or unruptured,
3. Aneurysm deemed by the attending neurointerventionalist to be acceptable candidates for endovascular embolization

Exclusion Criteria:

1) Patient / Treatment outside of the approved labeling, indications for use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2004-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To demonstrate performance of TRUFILL® DCS and TRUFILL DCS ORBIT™ Detachable Coils in the treatment of aneurysms | Between 3-6 months

SECONDARY OUTCOMES:
Adverse events and product complaints | Ongoing throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Bendok, M.D., Principal Investigator — Northwestern University
Locations (1):
- Kobe City General Hospital, Kobe, Japan

REFERENCES:
- [Background] Hirsch JA, Bendok BR, Paulsen RD, Cognard C, Campos J, Cronqvist M. Midterm clinical experience with a complex-shaped detachable platinum coil system for the treatment of cerebral aneurysms: Trufill DCS Orbit detachable coil system registry interim results. J Vasc Interv Radiol. 2007 Dec;18(12):1487-94. doi: 10.1016/j.jvir.2007.07.020. PMID 18057282